CLINICAL TRIAL: NCT07070986
Title: Randomized, Single-blind Pilot Study Assessing the Effect of Cutaneous RESonance Stimulation on SYMPAthetic and Parasympathetic Tone and Anxiety in Patients Admitted for Cardiac Surgery
Brief Title: Randomized, Single-blind Pilot Study Assessing the Effect of Cutaneous RESonance Stimulation SYMPAthetic and Parasympathetic Tone and Anxiety in Patients Admitted for Cardiac Surgery
Acronym: RESC SYMPA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1239
Record Dates: First submitted 2025-06-23; First posted 2025-07-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: Anxiety; Cardiac surgery; Pain; RESC
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CUTANEOUS RESONANCE STIMULATION (RESC): If randomized in the RESC group, interventional group, patient will receive a 20 minutes session of cutaneous resonance stimulation before his cardiac surgery according to a standardized protocol.
  Interventions: Procedure: RESC
- NON SPECIFIC CUTANEOUS STIMULATION (NSCS): If randomized in the NSCS group, control group, patient will receive a 20 minutes session of non-specific cutaneous stimulation before his cardiac surgery according to a standardized protocol.
  Interventions: Other: NSCS

INTERVENTIONS:
Procedure: RESC — If randomized in the RESC group, interventional group, patient will receive a 20 minutes session of cutaneous resonance stimulation before his cardiac surgery.
  He will be asked to respond to anxiety questionnaire STAI-E and to evaluate his anxiety on a visual analogue scale (VAS) at J-1 (day of inclusion), J0 (day of surgery), and J1 (the day after surgery).
  During the RESC session, LF/HF ratio, ANI, heart rate, respiratory rate, perfusion index and skin conductance will be monitored.
  Groups: CUTANEOUS RESONANCE STIMULATION (RESC)
Other: NSCS — If randomized in the NSCS group, interventional group, patient will receive a 20 minutes session of non-specific cutaneous stimulation before his cardiac surgery.
  He will be asked to respond to anxiety questionnaire STAI-E and to evaluate his anxiety on a visual analogue scale at J-1 (day of inclusion), J0 (day of surgery), and J1 (the day after surgery)
  During the NSCS session, LF/HF ratio, ANI, heart rate, respiratory rate, perfusion index and skin conductance will be monitored.
  Groups: NON SPECIFIC CUTANEOUS STIMULATION (NSCS)

SUMMARY:
Anxiety is a natural response to stress which peaks just before the surgery procedure. High levels of anxiety can increase postoperative pain and complications. Medicated anxiolysis is no longer recommended, in the absence of proven efficacy. Other interventions to prevent anxiety are required.

The autonomic nervous system (ANS), both sympathetic and parasympathetic, determines the response to stress. Anxiety interventions such as hypnosis, massage and relaxation work by modulating ANS tone. The ANS also modulates heart rate.

Anxiety can be measured by RR space, from which HRV, high-frequency (HF) and low-frequency (LF) are components respectively linked to the parasympathetic and sympathetic systems. The LF/HF ratio reflects sympathetic dominance if high, and parasympathetic dominance if low.

Cutaneous resonance stimulation (RESC) is a manual technique. RESC can diagnose and correct energy imbalances by skin stimulation between two points and thus act on anxiety.

We hypothesized that a preoperative RESC session would modify the sympathetic/parasympathetic balance and reduce anxiety in patients admitted for cardiac surgery, compared to patient receiving a sham RESC session: non-specific cutaneous stimulation (NSCS).

ELIGIBILITY:
Inclusion Criteria:

* Planned cardiac surgery with extracorporeal circulation
* Pre operatory anxiety : STAI-E score >30 or Visual Analogue Scale Anxiety >6

Exclusion Criteria:

* Urgent surgery
* Atrial fibrillation
* Impossibility to answer to STAI-E or VAS
* Use of alternative method
* Use of an alternative method other for anxiety before inclusion
* Absence of consent
* Pregnant, breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted for cardiac surgery with significant preoperative anxiety.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
LF/HF ratio variation compared between the groups | Between the beginning and the end of the RESC/NCS session (20 minutes)
  LF and HF will be monitored during the all RESC/NSCS.

SECONDARY OUTCOMES:
Skin conductance variation compared between the groups | Between the beginning and the end of the RESC/NCS session (20 minutes)
  Skin conductance will be monitored during the all RESC/NSC session.
Perfusion index variations compared between the groups. | Between the beginning and the end of the RESC/NCS session (20 minutes)
  Perfusion index ration will be monitored during the all RESC/NSC session.
Analgesia nociception index compared between the groups | Between the beginning and the end of the RESC/NCS session (20 minutes)
  Analgesia nociception index will be monitored during the all RESC/NSC session.
Anxiety compared between the groups | After de RESC/NCS session
  Anxiety will be assessed by visual analogue scale between 0 (no anxiety) and 10 (worst anxiety)
Morphine use post-surgery compared between the groups | Day 1
  Cumulative morphine used
Anxiety compared between the groups | After de RESC/NCS session
  Anxiety will be assessed by STAI-E
Heart rate variations compared between the groups. | Between the beginning and the end of the RESC/NCS session (20 minutes)
  Heart rate variation will be monitored during the all RESC/NSC session.
Blood pressure variations compared between the groups. | Between the beginning and the end of the RESC/NCS session (20 minutes)
  Blood pressure be monitored during the all RESC/NSC session.
Respiratory rate variations compared between the groups. | Between the beginning and the end of the RESC/NCS session (20 minutes)
  Respiratory rate will be monitored during the all RESC/NSC session.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitallouis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No